CLINICAL TRIAL: NCT03522688
Title: Impact of Dexmedetomidine on Acute Kidney Injury Following Living Donor Liver Transplantation: A Randomized Controlled Study
Brief Title: Impact of Dexmedetomidine on Acute Kidney Injury Following Living Donor Liver Transplantation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Jun-Gol Song, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DEX-LT
Record Dates: First submitted 2018-05-01; First posted 2018-05-11 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Acute Kidney Injury; Liver Diseases
Keywords: dexmedetomidine; acute kidney injury; liver transplantation
MeSH Terms: conditions — Acute Kidney Injury; Liver Diseases | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator): The control group was given normal saline by constant intravenous (IV) infusion at a rate of 0.4mcg/kg/hour
  Interventions: Drug: Normal saline
- treatment group (Active Comparator): The treatment group was given dexmedetomidine by constant intravenous (IV) infusion at a rate of 0.4mcg/kg/hour
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — The treatment group was given dexmedetomidine by constant intravenous (IV) infusion at a rate of 0.4mcg/kg/hour.
  Other Names: precedex
  Arms: treatment group
Drug: Normal saline — The control group was given normal saline by constant intravenous (IV) infusion at a rate of 0.4mcg/kg/hour
  Arms: control group

SUMMARY:
Acute kidney injury (AKI) following liver transplantation (LT) is associated with increased costs, morbidity, and mortality. Dexmedetomidine has known to have anti-inflammatory effect and has been shown to ameliorate IRI in several organs. However, the impact of Dexmedetomidine on AKI after LT is not determined yet. Therefore, this study aims to observe the renal protective effects of Dexmedetomidine after LT.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) following liver transplantation (LT) has shown a wide range of incidence between 17% and 95% and is associated with increased costs, morbidity, and mortality. The etiology of AKI after LT is multifactorial. Among these factors, renal ischemia-reperfusion injury (IRI) caused by perioperative renal hypoperfusion is considered as one of the most important independent risk factors and recent reports have indicated that IRI is associated with an inflammatory cascade. Dexmedetomidine which is a highly selective agonist of α2-adrenergic receptors has known have anti-inflammatory effect and has been shown to ameliorate IRI in several organs. However, the impact of Dexmedetomidine on AKI after LT is not determined yet. Therefore, this study aims to observe the renal protective effects of Dexmedetomidine after LT.

ELIGIBILITY:
Inclusion Criteria:

* living liver transplantation recipients

Exclusion Criteria:

* preoperative renal dysfunction
* dual living donor liver transplantation
* severe cerebral artery disease
* severe cardio-pulmonary disease

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2024-07-07 (Estimated)

PRIMARY OUTCOMES:
acute kidney injury | 7 days
  serum creatinine levels in postoperative 7 days

SECONDARY OUTCOMES:
lactate level | 3 days
  serial lactate level during operation and postoperative 3 days
delirium | postoperative day 7
  The incidence of delirium
early allograft dysfunction | postoperative day 7
  early allograft dysfunction
duration of mechanical ventilation | up to 1 year
  duration of mechanical ventilation (hours)
intensive care unit length of stay | up to 1 year
  intensive care unit length of stay (days)
hospital length of stay | up to 1 year
  hospital length of stay (days)
graft failure | 1 year
  recipient death or re-transplantation within 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Gol Song, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan medical center, Seoul, Songpa-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rimola A, Gavaler JS, Schade RR, el-Lankany S, Starzl TE, Van Thiel DH. Effects of renal impairment on liver transplantation. Gastroenterology. 1987 Jul;93(1):148-56. doi: 10.1016/0016-5085(87)90327-1. PMID 3556303
- [Background] Wyssusek KH, Keys AL, Yung J, Moloney ET, Sivalingam P, Paul SK. Evaluation of perioperative predictors of acute kidney injury post orthotopic liver transplantation. Anaesth Intensive Care. 2015 Nov;43(6):757-63. doi: 10.1177/0310057X1504300614. PMID 26603801
- [Background] Cho JS, Shim JK, Soh S, Kim MK, Kwak YL. Perioperative dexmedetomidine reduces the incidence and severity of acute kidney injury following valvular heart surgery. Kidney Int. 2016 Mar;89(3):693-700. doi: 10.1038/ki.2015.306. PMID 26444030
- [Background] Liu Y, Sheng B, Wang S, Lu F, Zhen J, Chen W. Dexmedetomidine prevents acute kidney injury after adult cardiac surgery: a meta-analysis of randomized controlled trials. BMC Anesthesiol. 2018 Jan 15;18(1):7. doi: 10.1186/s12871-018-0472-1. PMID 29334927

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-02): https://cdn.clinicaltrials.gov/large-docs/88/NCT03522688/Prot_SAP_000.pdf